CLINICAL TRIAL: NCT06708611
Title: A Crossover Study to Compare Natriuretic Effects of Extended Release Torsemide to Immediate Release Torsemide Over 12 Hours After Dosing in Patients with Heart Failure (EXTOR-HF)
Brief Title: A Crossover Study of Patients with HF to Compare Natriuretic Effects of IR Torsemide Vs. ER Torsemide Over 12 Hrs
Acronym: EXTOR-HF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Issues with recruitment
Sponsor: Sarfez Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAR065-324
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Torsemide

STUDY DESIGN:
Intervention Model Description: Double-blind, double-dummy, two-period, two arm, randomized, crossover clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Extended release torsemide (Experimental): Drug: Extended release torsemide 24 mg tablet. Subjects will receive oral dose of 24 mg extended release torsemide tablet and a placebo of 20 mg immediate release torsemide.
  Interventions: Drug: torsemide
- Immediate release torsemide (Active Comparator): Drug: Immediate release torsemide 20 mg tablet. Subjects will receive oral dose of 20 mg of immediate release torsemide and a placebo of 24 mg extended release torsemide.
  Interventions: Drug: torsemide

INTERVENTIONS:
Drug: torsemide — Extended release formulation of torsemide

SUMMARY:
This is a randomized double-blind crossover study of the patients with stable heart failure, who are taking a loop diuretic. During the study period, the participants' loop diuretics will be replaced by the equivalent dose of immediate release/extended release torsemide for one week. After a one week period, they will report to the site and will receive a single dose of either immediate release or extended release Torsemide. The sodium excretion will be measured for six hours after dosing and for an additional six hours after a high salt lunch.

DETAILED DESCRIPTION:
The goal of this randomized double-blind crossover study is to assess whether extended release torsemide has a better efficacy than immediate release torsemide to induce renal sodium excretion after a salty lunch in patients with heart failure. The study will address if:

* the amounts of excreted sodium in the urine during the 2- and 6-hours' time period after a morning dose of extended release torsemide is different from the amounts after the immediate release torsemide.
* the amounts of excreted sodium in the urine during the 2- and 6-hours' time period after a salty lunch, which will be consumed approximately 6 hours following a morning dose of extended release torsemide, is different from the amounts after the immediate release torsemide.
* the amount of excreted sodium in the urine during the 24 hours' time period after a salty lunch, which will be consumed approximately 6 hours following a morning dose of extended release torsemide, is different from the amount after the immediate release torsemide.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over the age of 18 years.
* Willing and able to sign the informed consent.
* A clinical diagnosis of chronic HF that is considered by patient's cardiologist/physician or an experienced clinician to be stable over the one-month period prior to randomization.
* Receiving oral furosemide (or equivalent doses of torsemide or bumetanide) for about 30 days prior to randomization.
* No anticipated changes in HF medications during the study period.
* Premenopausal women of child-bearing potential have a negative pregnancy test prior to beginning of the study and agree to use effective contraceptive methods during the study period

Exclusion Criteria:

* Requirement for a diuretic other than furosemide, bumetanide or torsemide except for spironolactone, eplerenone, finerenone, or SGLT2 inhibitors, at randomization and during the study.
* Myocardial infarction, stroke, transient ischemic attack, acute kidney injury or acute HF requiring admission to hospital within the last 30 days prior to randomization.
* Severe / symptomatic lung disease or respiratory symptoms distinct from HF.
* Urinary incontinence or inability to empty bladder.
* Uncontrolled diabetes mellitus or uncontrolled hypertension.
* Estimated GFR < 30 ml/min/1.72m2.
* History of flash pulmonary edema or amyloid cardiomyopathy.
* Female patients who are breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-03-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Cumulative Na+ excretion over 6 hours | 6 hours after lunch
  The primary outcome is the cumulative Na+ excretion over 6 hours after lunch.

SECONDARY OUTCOMES:
Fluid and Na+ excretion over the 6 hours | 6 hours after breakfast, 6 hours after lunch, and 24 hours]
  Fluid and Na+ excretion over the 6 hours after breakfast, 6 hours after lunch, and 24 hours after dosing.
Creatinine clearance | While in the study (approximately 2 weeks)
  Safety outcome
K+ excretion | While in the study (approximately 2 weeks)
  Safety outcome

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Shah, MD, Study Director — Safez Pharmaceuticals; Nayle A Ancares, MD, Principal Investigator — Future Life Clinical Trials
Locations (1):
- Future Life Clinical Trials, Miami, Florida, United States